CLINICAL TRIAL: NCT02981771
Title: The Effect of Exercise Training Programs - Stability and Coordination - On Static Balance, Dynamic Balance and Risk of Falls in Older Adults With Cardiovascular Disease
Brief Title: The Effect of Exercise Training Programs On Balance in Older Adults With CVD
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hillel Yaffe Medical Center (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: 0083-16-HYMC
Record Dates: First submitted 2016-11-29; First posted 2016-12-05 (Estimated); Last update posted 2018-10-17 (Actual); Status verified 2018-10

CONDITIONS: Aging; Cardiovascular Diseases
MeSH Terms: conditions — Cardiovascular Diseases

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- experiment (Experimental): A physical activity program that is based on balance and coordination exercises
  Interventions: Behavioral: Balance activity program
- control (Placebo Comparator): A physical activity program that is based on strength exercises
  Interventions: Behavioral: Strength activity program

INTERVENTIONS:
Behavioral: Balance activity program — Participants will take part in a biweekly, 12 week physical activity program that will include balance and coordination exercises
  Arms: experiment
Behavioral: Strength activity program — Participants will take part in a biweekly, 12 week physical activity program that will include traditional strength exercises
  Arms: control

SUMMARY:
Individuals of advanced age with cardiovascular disease are at higher risk of fall.The aim of this study is to explore the effect of specific exercise program based on balance and coordination on stability parameters

ELIGIBILITY:
Inclusion Criteria:

* Has Cardiovascular disease, under the supervision of a cardiologist
* Participates in a cardiovascular rehabilitation center
* Able to undergo physical activity for 60 minutes twice a week

Exclusion Criteria:

* All Other

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 31 (Actual)
Dates: Start 2017-02-08 (Actual); Primary Completion 2017-07-31 (Actual); Study Completion 2017-12-25 (Actual)

PRIMARY OUTCOMES:
Change in Balance ability - a composite outcome | 4 months
  In order to assess changes in balance ability, it will be measured with the following tests:
  Timed Get Up and Go , Balance Error Scoring System Test, Functional Reach Test, before and after the 12 week physical activity program and the difference will be compared

CONTACTS AND LOCATIONS:
Locations (1):
- Zinman College for Physical Education and Sport Sciences, Ramot Naftali, Israel